CLINICAL TRIAL: NCT02389855
Title: Laser Ablation in Stereotactic Neurosurgery
Brief Title: Laser Ablation in Stereotactic Neurosurgery (LAISE): NeuroBlate® Retrospective Registry
Status: Completed | Type: Observational
Sponsor: Monteris Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: LAISE
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Last update posted 2024-04-12 (Actual); Status verified 2021-08

CONDITIONS: Primary Brain Tumor
Keywords: Progression; Quality of Life
MeSH Terms: conditions — Brain Neoplasms; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: NeuroBlate® System Therapy

SUMMARY:
The NeuroBlate® System (NBS), is a minimally invasive robotic laser thermotherapy tool. It employs a pulsed surgical laser to deliver targeted energy to abnormal brain tissue caused by tumors and lesions. Since receiving FDA clearance in April 2013, the NBS has been used in nearly 300 procedures conducted at approximately 20 leading institutions across the United States. This post-market, multi-center retrospective study is designed to collect long-term follow-up data on patients who were treated previously with NBS.

ELIGIBILITY:
Inclusion Criteria:

* Patient was previously treated with NBS
* Patient is willing and able to provide informed consent and authorization for release of personal health information or IRB waiver is granted to collect study information without patient consent

Exclusion Criteria: There are no exclusion criteria for this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients previously treated with NBS (up to 300)
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2015-02; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Endpoint 1: Procedural Success Endpoint 2: Progression-Free Survival Endpoint 3: Overall Survival Endpoint 4: Karnofsky performance status | up to 24 months
  Retrospective data collection.

SECONDARY OUTCOMES:
Adverse Events | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Sujit Prabu, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center; Andrew Sloan, MD, PhD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (9):
- United States (9):
  - Yale University, New Haven, Connecticut
  - Kansas University Medical Center, Kansas City, Kansas
  - St. Luke's Hospital, Kansas City, Missouri
  - Washington University in St. Louis, St Louis, Missouri
  - Wake Forest, Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas